CLINICAL TRIAL: NCT06351891
Title: Efficacy and Safety of Bismuth Quadruple Therapy Containing Cefuroxime and Tetracycline as First-line Therapy for Eradicating Helicobacter Pylori in Patients Allergic to Penicillin: A Multicenter, Randomized Controlled Study
Brief Title: Efficacy and Safety of Bismuth Quadruple Therapy Containing Cefuroxime and Tetracycline as First-line Therapy for Eradicating Helicobacter Pylori in Patients Allergic to Penicillin
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHARE2402
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori Infection; Bismuth-containing quadruple therapy
MeSH Terms: interventions — Tetracycline; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14-day bismuth quadruple regimen containing cefuroxime and tetracycline (Experimental): 14-day bismuth quadruple regimen containing cefuroxime and tetracycline:Tegoprazan (50mg twice/day before breakfast and supper), Bismuth potassium citrate capsule (0.6g twice/day before breakfast and supper), Cefuroxime tablets (500mg twice/day after breakfast and supper), Tetracycline (500mg three times/day after three meals);14 days.
  Interventions: Drug: 14-day bismuth quadruple regimen containing cefuroxime and tetracycline
- 14-day bismuth quadruple regimen containing cefuroxime and levofloxacin (Active Comparator): 14-day bismuth quadruple regimen containing cefuroxime and levofloxacin:Tegoprazan (50mg twice/day before breakfast and supper), Bismuth potassium citrate capsule (0.6g twice/day before breakfast and supper), Cefuroxime tablets (500mg twice/day after breakfast and supper), Levofloxacin (500mg once/day after breakfast);14 days.
  Interventions: Drug: 14-day bismuth quadruple regimen containing cefuroxime and levofloxacin

INTERVENTIONS:
Drug: 14-day bismuth quadruple regimen containing cefuroxime and tetracycline — 14-day bismuth quadruple regimen containing cefuroxime and tetracycline:Tegoprazan 50mg bid, Bismuth potassium citrate capsules 0.6g bid,Cefuroxime tablets 500mg bid,Tetracycline 500mg tid,14 days.Evaluating the efficacy and safety of 14-Day bismuth quadruple therapy containing cefuroxime and tetracycline for Helicobacter pylori eradication.
  Arms: 14-day bismuth quadruple regimen containing cefuroxime and tetracycline
Drug: 14-day bismuth quadruple regimen containing cefuroxime and levofloxacin — 14-day bismuth quadruple regimen containing cefuroxime and levofloxacin:Tegoprazan 50mg bid, Bismuth potassium citrate capsules 0.6g bid,Cefuroxime tablets 500mg bid,Levofloxacin 500mg qd,14 days.
  Arms: 14-day bismuth quadruple regimen containing cefuroxime and levofloxacin

SUMMARY:
The researchers collected untreated H. pylori positive patients from outpatient clinics. Subjects were randomly assigned to receive either 14 days of bismuth quadruple therapy with cefuroxime and tetracycline or 14 days of bismuth quadruple therapy with cefuroxime and levofloxacin for Helicobacter pylori eradication. After 6 weeks of treatment, subjects underwent another 13C urea breath test. Eradication rates, adverse reaction rates and patient compliance were calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, regardless of gender.
2. History of penicillin allergy.
3. Helicobacter pylori infection.
4. Patients who have not previously received Helicobacter pylori eradication therapy.

Exclusion Criteria:

1. Medication history of bismuth and antibiotics within 4 weeks; PPIs and P-CABs within 2 weeks.
2. Serious underlying diseases, such as liver insufficiency, renal insufficiency, malignant tumors, etc.
3. Previous gastric or esophageal surgery.
4. History of allergy to test drugs.
5. Pregnant and lactating women and those unwilling to use contraception during the trial period.
6. Have other behaviors that may increase the risk such as alcohol and drug abuse.
7. Those unable to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | immediately after the procedure
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups.

SECONDARY OUTCOMES:
Rate of adverse reactions | immediately after the procedure
  Rate of adverse reactions
Patient compliance | immediately after the procedure
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Yueyue Li, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Wang H, Kong Q, Zhang Q, Zhang L, Li R, Zhang T, Guo L, Wang X, Li X, Zhao H, Liu F, Guo Y, Zhai Z, Li M, Yang X, Zuo X, Yang X, Li Y. Efficacy and Safety of Cefuroxime-Tetracycline-Containing Bismuth Quadruple Therapy for Helicobacter pylori Eradication in Penicillin-Allergic Patients: A Multicenter Randomized Controlled Trial. Helicobacter. 2025 Mar-Apr;30(2):e70033. doi: 10.1111/hel.70033. PMID 40237213